CLINICAL TRIAL: NCT05051293
Title: Comparison of the Concentration of Estrogen and Testosterone Ratio in Male Patients With Cirrhosis and Hypotension Compared to Male Cirrhosis Patients Without Hypotension
Brief Title: Comparison of the Concentration of Estrogen and Testosterone Ratio in Male Patients With Cirrhosis and Hypotension
Status: Withdrawn | Type: Observational
Why Stopped: Study will be changed from prospective to retrospective
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 097.HEP.2020.D
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-08

CONDITIONS: Hypotension; Cirrhosis
MeSH Terms: conditions — Hypotension; Fibrosis | interventions — methyl N-acetylsibirosaminide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- male cirrhotic with hypotension: Patients with cirrhosis have decreased spontaneous vascular resistance leading to hypotension.
  Interventions: Other: serum concentration of estrogen (E1 and E2) and testosterone ratio measurement
- male cirrhotic without hypotension: The concentration of estrogen in cirrhotic patients is thought to increase by fourfold compared to individuals without cirrhosis.
  Interventions: Other: serum concentration of estrogen (E1 and E2) and testosterone ratio measurement

INTERVENTIONS:
Other: serum concentration of estrogen (E1 and E2) and testosterone ratio measurement — To measure the serum concentration of estrogen (E1 and E2) and testosterone ratio in all male cirrhosis patients

SUMMARY:
Cirrhosis is an end stage in liver disease leading to replacement of normal liver tissue with regenerative nodules surrounded by fibrous bands in response to chronic liver injury. It is the eighth leading cause of death in the United States and the thirteenth leading cause of death globally. Patients with cirrhosis have decreased spontaneous vascular resistance leading to hypotension. The mechanism of hypotension in cirrhosis is thought to be a complex result of the presence of increased level of circulating vasodilators such a nitric oxide coupled with reduced resistance to vasoconstrictors and increased sensitivity to vasodilators.

DETAILED DESCRIPTION:
Another potential contributor to the development of hypotension in cirrhosis is thought to be due to the increased production of estrogen in males especially the estrone (E1) and estradiol (E2) concentration. The concentration of estrogen in cirrhotic patients is thought to increase by fourfold compared to individuals without cirrhosis. The increased estrogen concentration in cirrhosis patients results, in large part, from an increased peripheral conversion from androgens including testosterone. Previous studies have shown that increased estrogen concentration can cause a significant decrease in blood pressure in various cell, animal, and human models. Of note, estrogen has also been shown to enhance nitric oxide production in human beings.

ELIGIBILITY:
Inclusion Criteria:

* Male cirrhotic patients >18 years of age
* Patient must attend the outpatient clinic of the Liver Institute at Methodist Dallas Medical Center
* willing to provide informed consent to participate in the study

Exclusion Criteria:

* Patients with a history of cirrhosis <18 years of age
* Cirrhosis patients with active infection
* Cirrhosis patients with active gastrointestinal bleeding
* Cirrhosis patients on hormone replacement therapy testosterone
* Cirrhosis patients on any antihypertensive medications

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients attending the outpatient clinic of the Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-08-22 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2024-08-17 (Estimated)

PRIMARY OUTCOMES:
Serum estrogen (E1 and E2) levels | July to September 2021
  Measurement of serum estrogen (E1 and E2) levels in cirrhotic males
Serum testosterone levels | July to September 2021
  Measurement of serum testosterone levels in cirrhotic males

CONTACTS AND LOCATIONS:
Overall Officials: Mangesh Pagadala, MD, Principal Investigator — Methodist
Locations (1):
- Methodist Health System Clinical Research Institute, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ge PS, Runyon BA. Treatment of Patients with Cirrhosis. N Engl J Med. 2016 Nov 24;375(21):2104-5. doi: 10.1056/NEJMc1612334. No abstract available. PMID 28121086
- [Background] Iwakiri Y, Groszmann RJ. The hyperdynamic circulation of chronic liver diseases: from the patient to the molecule. Hepatology. 2006 Feb;43(2 Suppl 1):S121-31. doi: 10.1002/hep.20993. PMID 16447289
- [Background] Cavanaugh J, Niewoehner CB, Nuttall FQ. Gynecomastia and cirrhosis of the liver. Arch Intern Med. 1990 Mar;150(3):563-5. PMID 2310274
- [Background] Gordon GG, Olivo J, Rafil F, Southren AL. Conversion of androgens to estrogens in cirrhosis of the liver. J Clin Endocrinol Metab. 1975 Jun;40(6):1018-26. doi: 10.1210/jcem-40-6-1018. PMID 1133151
- [Background] Seely EW, Walsh BW, Gerhard MD, Williams GH. Estradiol with or without progesterone and ambulatory blood pressure in postmenopausal women. Hypertension. 1999 May;33(5):1190-4. doi: 10.1161/01.hyp.33.5.1190. PMID 10334810